CLINICAL TRIAL: NCT02301520
Title: Vitamin D Deficiency, Iodine Deficiency and Lead Levels in Haitian Infants and Children.
Brief Title: Vitamin D, Iodine, and Lead Levels in Haitian Infants and Children.
Acronym: Haiti
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Fondation Haitienne de Diabete et de Maladies Cardiovasculaires (FHADIMAC) (Unknown); Kay Mackenson Clinic, Inc. (Other)
Responsible Party: Principal Investigator, Julia Von Oettingen, Fellow in Pediatric Endocrinology, Boston Children's Hospital
Other Study IDs: Haitistudy
Record Dates: First submitted 2014-11-23; First posted 2014-11-26 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Vitamin D Deficiency; Iodine Deficiency; Hypothyroidism; Rickets; Lead Intoxication
Keywords: Vitamin D; Iodine; Lead; Thyroid function; point-of-care test
MeSH Terms: conditions — Vitamin D Deficiency; Hypothyroidism; Rickets; Lead Poisoning

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Vitamin D deficiency is common worldwide, including in infants and children, and rickets remains a public health concern in many developing countries. The vitamin D status and prevalence of vitamin D deficiency in the Haitian population has not been studied. There is currently no approved point-of-care testing device for vitamin D deficiency. Iodine deficiency and resulting hypothyroidism is the leading cause of preventable neuro-developmental delay and cognitive impairment worldwide. Young infants and children are especially susceptible to sequelae of disruption in thyroid function given the dependence of the developing brain on sufficient levels of thyroid hormone. Perchlorate and thiocyanate have been described as potential environmental disrupters of thyroid function. Lead intoxication is a significant cause of disease throughout the world. Millions of people have suffered the effects of lead poisoning. Although most developed countries have taken drastic measures to limit the environmental lead levels, many countries in the developing world have not been able to address, or even assess, the problem.

Our objectives are to study the following three components in 300 Haitian children between 9 months and 6 years of age in three different geographical areas of Haiti: 1) Vitamin D status and prevalence of rickets, environmental factors associated with low vitamin D levels, and the accuracy and efficacy of a vitamin D point-of-care testing (POCT) device for the screening of vitamin D insufficiency. 2) Iodine status and thyroid function, and environmental disruptors such as perchlorate and thiocyanate as potential risk factors for abnormal thyroid function. 3) Lead levels and the extent of childhood lead poisoning.

DETAILED DESCRIPTION:
BACKGROUND:

1. Vitamin D Deficiency

   Vitamin D deficiency is common in the United States and worldwide, including in infants and children 1,2. Moderate to severe deficiency in children can manifest as rickets, a skeletal disease which results from a failure of mineralization of developing bones and cartilage. In most industrialized countries, infantile vitamin D supplementation represents the standard of care and has lead to a dramatic reduction in the incidence of rickets. However, in many developing countries, rickets remains a public health problem 3.In addition, recent literature indicates that there may be a resurgence of rickets even in industrialized countries 4, especially among immigrant populations 5. Potential extraskeletal effects of vitamin D deficiency are also being increasingly recognized, including an increased susceptibility to type 1 diabetes, insulin resistance and the metabolic syndrome, pulmonary disease such as asthma, pneumonia and tuberculosis, and possible modulation of the innate immune system 6.

   Growing children with severe vitamin D deficiency, most commonly defined as serum 25-hydroxy-vitamin D (25OHD) levels less than 8 ng/ml, are at greatest risk for rickets and should undergo a diagnostic evaluation. When physical exam findings such as bowing of weight-bearing extremities, rachitic rosary, or frontal bossing are not evident, the level of serum alkaline phosphatase as an indicator for increased bone turnover and calcium mobilization from bone can be used as a screening test 4,7. X-rays of knees and wrists are typically obtained to confirm the diagnosis and establish a baseline for follow up.

   The vitamin D status and prevalence of vitamin D deficiency in the Haitian population has not been studied. The prevalence of rickets is also unknown. Two studies conducted in Puerto Rican children 8 and in newly immigrated adults of Caribbean background 9 found prevalence rates of 47% and 59%, respectively, suggesting the possibility of moderate to high prevalence rates in Haiti.

   The best indicator to assess vitamin D status is the 25OHD metabolite, the major circulating form of vitamin D 10. There is no international consensus on the definition of vitamin D deficiency. The Institute of Medicine defines deficiency as a 25OHD < 20ng/mL and suggests levels be maintained above this threshold for healthy children and adolescents 11. The Endocrine Society recommendations were aimed at children and adults with chronic conditions placing them at risk for a low bone mass and/or vitamin D deficiency, and recommend using a level below 30 ng/mL (80 nmol/L) to define insufficiency and below 20 ng/mL (50 nmol/L) to define deficiency 6. The Endocrine Society treatment guideline for vitamin D deficiency for children 0-18 years suggests administering oral vitamin D3 2000 IU daily or 50,000 IU weekly for 6 weeks, followed by an age-appropriate maintenance dose.

   In resource limited settings, laboratory facilities for vitamin D testing are frequently unavailable. A point-of-care testing method would greatly facilitate screening for vitamin D deficiency and insufficiency. The test 4D is a novel point-of-care test device that is not yet FDA licensed. Only manufacturer based information on test accuracy are currently available. The device has not been tested in children (package insert is attached to this protocol).
2. Iodine Deficiency

   Iodine deficiency and resulting hypothyroidism is the leading cause of preventable neuro-developmental delay and cognitive impairment worldwide. Young infants and children are especially susceptible to sequelae of disruption in thyroid function given the dependence of the developing brain on sufficient levels of thyroid hormone.

   Urinary iodine has been established as the gold standard for the assessment of iodine status12. Values of 100-199 mcg/L are considered optimal, whereas levels <100 mcg/L, <50 mcg/dL and <20 mcg/dL define mild, moderate and severe iodine deficiency, respectively. On the other hand, the risk of iodine induced hyperthyroidism increases when levels rise to 200 mcg/dl and above, and risk of adverse health consequences increases with levels exceeding 300 mcg/L12. Perchlorate and thiocyanate are environmental chemicals known to inhibit the sodium-iodine symporter when administered at pharmacologic doses. This leads to interference with normal thyroidal iodine uptake and results in decreased thyroid hormone production13,14. Both chemicals do not undergo significant metabolism and can be readily detected in the urine. The effect of environmental exposure to either is thought to be dependent on adequate iodine, and should thus be assessed concurrent with urinary iodine status14.

   Studies assessing the iodine status in Haiti are few in number and have mainly included school-age children and adults. Three studies in school-aged children conducted between 1996 and 2002 have found moderate to severe iodine deficiency, with urinary iodine levels ranging between 38.8 and 43.4 mcg/dL15-17, regardless of whether children from coastal15,16 or mountainous regions17 were surveyed. One study found elevated TSH values >5 mU/L in 78.5% of participants15. A more recent study conducted in 2008 examined 88 subjects between ages 2 and 72 years, and found a similar median urinary iodine concentration18. Overall, between 60 and over 90% of the Haitian population may be iodine deficient17-19, with up to 20% falling into the range of severe deficiency18. Based on WHO data from 2005 to 2006, only 3% of households are consuming adequately iodized salt19. No studies have been conducted in infants and children under the age of 5 years..

   The proposed study will be the first to assess the iodine status of Haitian infants and young children. The study will be conducted in 3 different geographical areas of the country, including an urban setting (Port-au-Prince), a mountainous region (Central Plateau), and a coastal area (Saint Marc) in an attempt to differentiate between areas where iodine deficiency is more likely (Central Plateau) from those were it is less likely (Saint Marc). For the first time, urinary iodine concentration in young children will be obtained along with a clinical goiter assessment, concentrations of urinary perchlorate and thiocyanate, as well as thyroid function studies (thyroid stimulating hormone and free thyroxine).

   Confirmation of iodine deficiency may have significant public health implications for one of the most vulnerable populations: infants and young children. Improving their access to iodized salt and/or iodine supplementation could have a major impact on reducing the number of children (and future adults) with hypothyroidism-related mental retardation. The study results may raise awareness of medical providers with regards to the problem of iodine deficiency and related hypothyroidism, and may provide an incentive to test children for hypothyroidism. There may be other major clinical implications, including the ability to detect and treat affected children, and improve their prognosis with regards to cognitive impairment. On a larger scale, depending on the magnitude of the problem, the study findings may underline the need to assess iodine deficiency and hypothyroidism in even younger infants, including newborns. Results may further obviate the need for a newborn screening program for hypothyroidism in Haiti.
3. Lead Intoxication

Lead intoxication is a significant cause of disease throughout the world. Millions of people have suffered the effects of lead poisoning. Although most developed countries have taken drastic measures to limit the environmental lead levels, many countries in the developing world have not been able to address, or even assess, the problem.

Lead poisoning is a medical condition caused by increased levels of lead in the body. Lead is a highly toxic heavy metal environmental toxicant and nerve poison that can contribute to the destruction of many developmental functions by interfering with a variety of body processes. Due to its insidious nature, lead causes subtle and sometimes unnoticeable effects in children. Even low levels of lead exposure among children can be associated with developmental problems including impaired cognitive function, reduced intelligence, impaired hearing, reduced stature or damage to the bone marrow 20,21. Lead poisoning can cause severe toxicities including convulsions, coma, and death 22. In the United States, the Centers for Disease Control and Prevention (CDC) define an elevated child BLL as ≥ 10 µg/dL. At this BLL, the CDC has given permission to initiate public health actions. Additionally, the CDC has also recommended that children with BLLs ≥ 45 µg/dL receive intensive medical management and chelation therapy 23 to prevent irreversible damage to the child.

Among developing countries, major sources of childhood lead poisoning include lead mining and smelting, paint, leaded gasoline, battery recycling, and traditional medicines 24,25 Despite the abundance of lead containing materials available in these developing countries, there are still a limited number of studies that have actually documented environmental lead contamination. Even with documented cases, information is further limited to adults living in small-scale gold ore-processing communities 26-29. Despite the many advances of treatment of lead poisoning in the US, there is still a paucity of information for childhood lead poisoning in the developing world.

The proposed study will document lead levels in the pediatric population in three different regions of Haiti. Data obtained from this study may lead to clinically relevant prognostic, diagnostic or therapeutic modalities. This information may further be used to implement or even eradicate lead as a public health hazard.

STUDY OBJECTIVES

Our objectives are to study the following three components in 300 Haitian children between 9 months and 6 years of age in three different geographical areas of Haiti: 1) Vitamin D status and prevalence of rickets, environmental factors associated with low vitamin D levels, and the accuracy and efficacy of a vitamin D point-of-care testing (POCT) device for the screening of vitamin D insufficiency. 2) Iodine status and thyroid function, and environmental disruptors such as perchlorate and thiocyanate as potential risk factors for abnormal thyroid function. 3) Lead levels and the extent of childhood lead poisoning.

Aim 1: To determine the proportion of children with vitamin D insufficiency, deficiency and severe deficiency, as defined by serum 25-hydroxyvitamin D (25OHD) levels <30ng/ml, <20 ng/ml, and <10 ng/ml, respectively.

Aim 2: To determine the proportion of children at high risk for rickets as defined by vitamin D deficiency and elevations in alkaline phosphatase.

Aim 3: To determine the extent to which dietary vitamin D intake and sun exposure are related to serum 25OHD levels.

Aim 4: To correlate the results from a vitamin D POCT device with serum 25OHD levels.

Aim 5: To determine the prevalence of iodine deficiency. Aim 6: To assess the subjects' thyroid function (TSH and free T4). Aim 7: To screen for urinary presence of two potential environmental disruptors of thyroid hormone production.

Aim 8: To determine the correlation of abnormal thyroid function, geographical area, and presence of urinary perchlorate and thiocyanate with iodine status.

Aim 9: To determine the mean and range of blood lead levels (BLL). Aim 10: To determine the proportion of children with a blood lead level (BLL) ≥ 10 µg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Haitian ethnicity
* Age between nine months and six years

Exclusion Criteria:

* Presence of a chronic medical condition other than malnutrition
* Residence outside of Haiti (i.e. visiting children who usually live abroad).

Ages: 9 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants and young children, recruited from participating local churches in three different geographical areas of Haiti, including in the capital Port-au-Prince, a mountainous region, and a coastal region.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
serum 25OHD levels | Baseline
  Measure serum 25OHD levels, including the proportion of children found to be vitamin D insufficient, deficient and severely deficient.
urinary iodine levels | Baseline
  Urinary iodine levels, including the proportion of children found to be iodine deficient
serum lead levels | Baseline
  Serum lead levels in Haitian infants and children

SECONDARY OUTCOMES:
Number of children found to have elevated alkaline phosphatase levels | Baseline
  The number of vitamin D deficient children found to have elevated alkaline phosphatase levels (as a proxy for vitamin D deficient rickets)
Dietary and sun exposure effect on vitamin D level | Baseline
  to measure the influence of dietary vitamin D intake and sun exposure on vitamin D levels.
Determine the accuracy of the POCT device | Baseline
  The 25OHD levels were measured via serum and POCT device to compare accuracy of the POCT device.
Goiter and abnormal thyroid function tests | Baseline
  The number of children found to have goiters and/or abnormal thyroid function tests
Environmental disruptors of thyroid function | Baseline
  Number of children with elevated levels of urinary perchlorate and/or thiocyanate
Lead intoxication | Baseline
  Evaluation of the extent of childhood lead poisoning using the CDC definition of lead poisoning, (BLL) ≥ 10 µg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Julia Von Oettingen, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- Haiti (2):
  - Kay Mackenson Clinic, Pierre Payen
  - FHADIMAC, Port-au-Prince

REFERENCES:
- [Background] Gordon CM, Feldman HA, Sinclair L, Williams AL, Kleinman PK, Perez-Rossello J, Cox JE. Prevalence of vitamin D deficiency among healthy infants and toddlers. Arch Pediatr Adolesc Med. 2008 Jun;162(6):505-12. doi: 10.1001/archpedi.162.6.505. PMID 18524739
- [Background] Misra M, Pacaud D, Petryk A, Collett-Solberg PF, Kappy M; Drug and Therapeutics Committee of the Lawson Wilkins Pediatric Endocrine Society. Vitamin D deficiency in children and its management: review of current knowledge and recommendations. Pediatrics. 2008 Aug;122(2):398-417. doi: 10.1542/peds.2007-1894. PMID 18676559
- [Background] Weisberg P, Scanlon KS, Li R, Cogswell ME. Nutritional rickets among children in the United States: review of cases reported between 1986 and 2003. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1697S-705S. doi: 10.1093/ajcn/80.6.1697S. PMID 15585790
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Holick MF. Vitamin D deficiency. N Engl J Med. 2007 Jul 19;357(3):266-81. doi: 10.1056/NEJMra070553. No abstract available. PMID 17634462
- [Background] Taylor JA, Richter M, Done S, Feldman KW. The utility of alkaline phosphatase measurement as a screening test for rickets in breast-fed infants and toddlers: a study from the puget sound pediatric research network. Clin Pediatr (Phila). 2010 Dec;49(12):1103-10. doi: 10.1177/0009922810376993. Epub 2010 Aug 19. PMID 20724326
- [Background] Mughal MZ. Rickets. Curr Osteoporos Rep. 2011 Dec;9(4):291-9. doi: 10.1007/s11914-011-0081-0. PMID 21968816
- [Background] Brehm JM, Acosta-Perez E, Klei L, Roeder K, Barmada M, Boutaoui N, Forno E, Kelly R, Paul K, Sylvia J, Litonjua AA, Cabana M, Alvarez M, Colon-Semidey A, Canino G, Celedon JC. Vitamin D insufficiency and severe asthma exacerbations in Puerto Rican children. Am J Respir Crit Care Med. 2012 Jul 15;186(2):140-6. doi: 10.1164/rccm.201203-0431OC. Epub 2012 May 31. PMID 22652028
- [Background] Penrose K, Hunter Adams J, Nguyen T, Cochran J, Geltman PL. Vitamin D deficiency among newly resettled refugees in Massachusetts. J Immigr Minor Health. 2012 Dec;14(6):941-8. doi: 10.1007/s10903-012-9603-9. PMID 22411495
- [Background] Shaw NJ, Mughal MZ. Vitamin D and child health: part 2 (extraskeletal and other aspects). Arch Dis Child. 2013 May;98(5):368-72. doi: 10.1136/archdischild-2012-302585. Epub 2013 Mar 14. PMID 23493188
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] de Benoist B, McLean E, Andersson M, Rogers L. Iodine deficiency in 2007: global progress since 2003. Food Nutr Bull. 2008 Sep;29(3):195-202. doi: 10.1177/156482650802900305. PMID 18947032
- [Background] Leung AM, Pearce EN, Braverman LE. Perchlorate, iodine and the thyroid. Best Pract Res Clin Endocrinol Metab. 2010 Feb;24(1):133-41. doi: 10.1016/j.beem.2009.08.009. PMID 20172477
- [Background] Pearce EN, Braverman LE. Environmental pollutants and the thyroid. Best Pract Res Clin Endocrinol Metab. 2009 Dec;23(6):801-13. doi: 10.1016/j.beem.2009.06.003. PMID 19942155
- [Background] Beach MJ, Streit TG, Houston R, May WA, Addiss DG, Lammie PJ. Short report: documentation of iodine deficiency in Haitian schoolchildren: implication for lymphatic filariasis elimination in Haiti. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2):56-7. doi: 10.4269/ajtmh.2001.64.56. PMID 11425163
- [Background] Freeman AR, Lammie PJ, Houston R, LaPointe MD, Streit TG, Jooste PL, Brissau JM, Lafontant JG, Addiss DG. A community-based trial for the control of lymphatic filariasis and iodine deficiency using salt fortified with diethylcarbamazine and iodine. Am J Trop Med Hyg. 2001 Dec;65(6):865-71. doi: 10.4269/ajtmh.2001.65.865. PMID 11791989
- [Background] Pilliod, K. Iodine Deficiency in Haiti : 16, i-43 (2003).
- [Background] Tenpenny KE, Trent CJ, Sutherland PA, Van Middlesworth L, Williams-Cleaves B, Braverman LE. Evidence of endemic goiter and iodine deficiency in a mountainous area of Haiti. Endocr Pract. 2009 May-Jun;15(4):298-301. doi: 10.4158/EP08330.ORR1. PMID 19454392
- [Background] World Health Organization. Assessment of iodine deficiency disorders and monitoring their elimination. WHO 2001.
- [Background] Canfield RL, Henderson CR Jr, Cory-Slechta DA, Cox C, Jusko TA, Lanphear BP. Intellectual impairment in children with blood lead concentrations below 10 microg per deciliter. N Engl J Med. 2003 Apr 17;348(16):1517-26. doi: 10.1056/NEJMoa022848. PMID 12700371
- [Background] Jusko TA, Henderson CR, Lanphear BP, Cory-Slechta DA, Parsons PJ, Canfield RL. Blood lead concentrations < 10 microg/dL and child intelligence at 6 years of age. Environ Health Perspect. 2008 Feb;116(2):243-8. doi: 10.1289/ehp.10424. PMID 18288325
- [Background] Needleman H. Lead poisoning. Annu Rev Med. 2004;55:209-22. doi: 10.1146/annurev.med.55.091902.103653. PMID 14746518
- [Background] Managing Elevated Blood Lead Levels among Young Children: Recommendations from the Advisory Committee on Childhood. Centers Dis. Control Prev. at <http://www.cdc.gov/nceh/lead/casemanagement/casemanage_main.htm>
- [Background] Falk H. International environmental health for the pediatrician: case study of lead poisoning. Pediatrics. 2003 Jul;112(1 Pt 2):259-64. PMID 12837919
- [Background] Meyer PA, Brown MJ, Falk H. Global approach to reducing lead exposure and poisoning. Mutat Res. 2008 Jul-Aug;659(1-2):166-75. doi: 10.1016/j.mrrev.2008.03.003. Epub 2008 Mar 20. PMID 18436472
- [Background] Appleton, J. D., Williams, T. M., Orbea, H. & Carrasco, M. Fluvial Contamination Associated with Artisanal Gold Mining in the Ponce Enríquez, Portovelo-Zaruma and Nambija Areas, Ecuador. Water. Air. Soil Pollut. 131, 19-39 (2001).
- [Background] Odumo OB, Mustapha AO, Patel JP, Angeyo HK. Multielemental analysis of Migori (Southwest, Kenya) artisanal gold mine ores and sediments by EDX-ray fluorescence technique: implications of occupational exposure and environmental impact. Bull Environ Contam Toxicol. 2011 May;86(5):484-9. doi: 10.1007/s00128-011-0242-y. Epub 2011 Mar 20. PMID 21424574
- [Background] Betancourt, O., Narváez, A. & Roulet, M. Small-scale Gold Mining in the Puyango River Basin,Southern Ecuador: A Study of Environmental Impacts andHuman Exposures. Ecohealth 2, 323-332 (2005).
- [Background] Ogola, J. S., Mitullah, W. V. & Omulo, M. A. Impact of Gold mining on the Environment and Human Health: A Case Study in the Migori Gold Belt, Kenya. Environ. Geochem. Health 24, 141-157 (2002).
- [Background] Putman MS, Pitts SA, Milliren CE, Feldman HA, Reinold K, Gordon CM. A randomized clinical trial of vitamin D supplementation in healthy adolescents. J Adolesc Health. 2013 May;52(5):592-8. doi: 10.1016/j.jadohealth.2012.10.270. Epub 2012 Dec 23. PMID 23608721
- [Background] Salamone LM, Dallal GE, Zantos D, Makrauer F, Dawson-Hughes B. Contributions of vitamin D intake and seasonal sunlight exposure to plasma 25-hydroxyvitamin D concentration in elderly women. Am J Clin Nutr. 1994 Jan;59(1):80-6. doi: 10.1093/ajcn/59.1.80. PMID 8279408
- [Background] Valentin-Blasini L, Mauldin JP, Maple D, Blount BC. Analysis of perchlorate in human urine using ion chromatography and electrospray tandem mass spectrometry. Anal Chem. 2005 Apr 15;77(8):2475-81. doi: 10.1021/ac048365f. PMID 15828783
- [Derived] von Oettingen JE, Brathwaite TD, Carpenter C, Bonnell R, He X, Braverman LE, Pearce EN, Larco P, Larco NC, Jean-Baptiste E, Brown RS. Population Survey of Iodine Deficiency and Environmental Disruptors of Thyroid Function in Young Children in Haiti. J Clin Endocrinol Metab. 2017 Feb 1;102(2):644-651. doi: 10.1210/jc.2016-2630. PMID 27768855